CLINICAL TRIAL: NCT05175287
Title: Risk of Obstructive Sleep Apnea and Traffic Accidents Among Bus Drivers in Ecuador: is There a Significant Association
Brief Title: OSA (oRisk of Obstructive Sleep Apnea and Traffic Accidents Among Bus Drivers in Ecuador: is There a Significant Association
Status: Completed | Type: Observational
Sponsor: Respiralab (Other)
Collaborators: Universidad de Especialidades Espíritu Santo (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2021-MED-002
Record Dates: First submitted 2021-12-14; First posted 2022-01-03 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Sleep Apnea, Obstructive
Keywords: Sleep apnea; daytime sleepiness; accidents; bus drivers
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes; Disorders of Excessive Somnolence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Our study aims to determine the frequency of individuals at high risk of obstructive sleep apnea, and excessive daytime sleepiness, as well as any potential association between these conditions and traffic accidents among a sample of Ecuadorian bus drivers.

DETAILED DESCRIPTION:
We conducted a cross-sectional study from September 2019 to January 2020 among 340 male professional bus drivers in the city of Guayaquil, Ecuador. To be included in the study, participants were required to be male, have an unexpired professional driver's license, as well as being currently enrolled at any local transformational company. Individuals who did not met the inclusion criteria, or who declined voluntary participation were excluded from the study. We screened 340 male professional bus drivers whose mean age was 44.3. We analyzed demographic and clinical variables including age, educational level, associated comorbidities (hypertension and diabetes), years as a professional driver, and number of accidents and near-accidents while working. Accidents were defined as a collision involving the vehicle in which the participant was the driver and another vehicle or stationary obstruction. Near-accidents were defined as unplanned events involving the driver that did not result in injury but had the potential to do so. We used STOP questionnaire to assess four questions related to snoring, tiredness during daytime, observed apnea, and high blood pressure (STOP), and the Bang aspect for screening BMI ≥ 35, age ≥ 50, neck circumference > 40 cm and male gender. Also, we used Epworth Sleepiness Scale (ESS) to assess excessive daytime sleepiness (EDS).

ELIGIBILITY:
Inclusion Criteria:

* Male
* Have an unexpired professional driver's license
* Being currently enrolled at any local transformational company

Exclusion Criteria:

* Not meeting inclusion criteria
* Declined voluntary participation

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 340 male professional bus drivers whose mean age was 44.3 in the city of Guayaquil, Ecuador.
Sampling Method: Non-Probability Sample
Enrollment: 340 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-02-15 (Actual)

PRIMARY OUTCOMES:
Obstructive sleep apnea | 4 months
  STOP-Bang questionnaire: assesses four questions related to snoring, tiredness during daytime, observed apnea, and high blood pressure (STOP), while the Bang aspect screens for a BMI ≥ 35, age ≥ 50, neck circumference > 40 cm and male gender.

SECONDARY OUTCOMES:
Excessive daytime sleepiness (EDS) | 4 months
  Epworth Sleepiness Scale (ESS): self-administered questionnaire, with 8 questions in which individuals are asked to rate the likelihood of falling asleep while engaged in different activities using a 4-point scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Respiralab Research Group, Guayaquil, Guayas, Ecuador